CLINICAL TRIAL: NCT01794156
Title: Evaluation of a Cognitive Therapy (Inference-based-therapy) for the Treatment of Obsessional Compulsive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre de Recherche de l'Institut Universitaire en santé Mentale de Montréal (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Frederick Aardema, Ph. D., Centre de Recherche de l'Institut Universitaire en santé Mentale de Montréal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 119587
Record Dates: First submitted 2013-02-07; First posted 2013-02-18 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Obsessive Compulsive Disorder
Keywords: Inference-based therapy; Cognitive behavior therapy; Obsessive compulsive disorder; Randomized clinical trial
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cognitive Behavioral Therapy; Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cognitive behavior therapy (Active Comparator): 1. The cognitive-behavioral model is presented and individualized.
  2. Cognitive correction: beliefs are addressed by explaining their roles in maintaining cognitive biases. Next, clients are trained to identify and to challenge their key beliefs
  3. Exposure and response prevention (ERP) using imaginal and in vivo exposure and to both over and covert neutralization is implemented according to hierarchies developed following the individual assessment. Extended periods of exposure permits emotional discomfort to dissipate.
  4. Combined phase: continues ERP while making explicit links to the cognitive targets.
  5. Relapse prevention included a written individualized guide to encourage the maintenance of treatment gains. Self-directed ERP continues.
  Interventions: Behavioral: Cognitive behavior therapy
- Mindfulness-based stress reduction (MBSR) (Active Comparator): The entire intervention is based on systematic and intensive training in MBSR following Santorelli and Kabat-Zinn and their applications to everyday life. The program is divided in 8 consecutive blocks with daily homework in mindfulness-based stress reduction skills. The main activity of MBSR is a cognitive and intervention-based process characterized by self-regulation of attention to the present moment and an open and accepting orientation towards one's experience.
  Interventions: Behavioral: Mindfulness-based stress reduction
- Inference-based therapy (Experimental): The inference-based therapy will be delivered in 10-step
  The client will:
  * learn that the compulsions, anxiety and discomfort are driven by an initial obsessional doubt
  * learn why this doubt is 100% irrelevant here and now
  * learn the inferential confusion process
  * have to recognize that the doubt originates from him/her
  * have to identify/describe the narrative leading him/her to the doubt
  * have to identify the cross-over point when he/she leaves reality
  * learn to be aware of the reasoning devices
  * learn how personal themes dictate the idiosyncratic nature of the person's obsession
  * explore and reinforced an alternative self-view
  * be trained to use properly his/her senses in the face of obsessional triggers situations
  Interventions: Behavioral: Inference-based therapy

INTERVENTIONS:
Behavioral: Cognitive behavior therapy
  Arms: Cognitive behavior therapy
Behavioral: Mindfulness-based stress reduction
  Arms: Mindfulness-based stress reduction (MBSR)
Behavioral: Inference-based therapy
  Arms: Inference-based therapy

SUMMARY:
Obsessional compulsive disorder (OCD) is a very debilitating psychiatric problem which affects around one million Canadians and their families. Obsessions are intense preoccupations about bad, harmful, dangerous, shocking or unlucky events which 'may' occur and which drive sufferers to perform time consuming and distressing compulsive rituals to prevent the possible event occurring. The current psychological treatment of choice is cognitive behavior (CBT) therapy which focuses on treating OCD by reducing obsessional anxiety about the likelihood and the consequences of the preoccupying event. A rival cognitive model termed the inference-based therapy (IBT), developed by the principal investigator and co-workers, considers that the OCD begins with the initial doubting inference 'maybe something is wrong' and focuses on changing the reasoning behind this doubting inference which often trumps the common sense conviction that there is no reason to doubt. This clinical trial randomly allocates participants to either IBT or CBT treatment condition or to a third generic mindfulness condition. The latter condition is a non-specific meditational-based training which has shown evidence of reducing stress and anxiety across a number of psychiatric problems including OCD. Two hundred and forty people will be recruited over a 5-year period from two principal sites (Montreal and Gatineau/Ottawa) with which the principal investigator and co-investigators have clinical links. Therapy will be administered by trained professionals following a treatment manual specific to each approach. The therapy will last a maximum of six months or until the point when the person achieves a non-clinical status. The patients will be assessed pre, post, and at six months following treatment on standard evaluation instruments as well as on subjective measures. We expect the IBT to be superior in terms of number of participants responding to treatment, rapidity of improvement and gains at follow-up.

DETAILED DESCRIPTION:
Obsessive compulsive disorder (OCD) affects 1-3% of the population and is the fourth most common mental disorder. It is characterized by a preoccupying obsessional doubt that harm, illness, disorder or bad luck, will occur if compulsive actions are not carried out to neutralize the risk. Treatments of choice include pharmacotherapy and cognitive behavior therapy (CBT) either alone or in combination. Although these interventions are clinically effective, they usually do not reduce the obsessions to a sub-clinical level. There is a risk of relapse and even so a sizeable minority of people with OCD refuse or abandon treatment, and some specific subtypes of OCD show no or minimal response. CBT-as-usual, involves principally the administration of exposure and response prevention (E/RP). A cognitive psycho-education element may by added in line with current cognitive thinking that it is the appraisal the person attributes to the initial intrusive thought with engenders obsessional distress. Such cognitive treatment will focus on modifying the anxiety and beliefs about consequences following on from the initial obsessional preoccupation. A competing cognitive model termed the inference-based approach (IBA) developed by the principal investigator and co-workers offers an account of obsessions which focuses on the reasoning producing the initial obsessional doubt as the source of the OCD. In this model the obsessing begins at the point where the person crosses over from reality into the initial obsessional doubt since the doubt is not based on real perception but on a subjective narrative misleading the person to infer doubt where no doubt is required. Over the last 10 years, experimental, clinical and psychometric research studies (independently replicated) have supported the essential claims of the IBA and have led to development of inference-based therapy (IBT). A small scale randomized clinical trial, and clinical case studies have established IBT as a 'promising' intervention (according to American Psychological Association criteria) and shown that IBT seems to offer advantages over conventional CBT, particularly for treatment-resistant cases who over-invest in their obsessional convictions. The current randomized clinical trial will compare IBT to CBT as usual, and to a third active control condition of mindfulness. Mindfulness is a generic treatment shown effective in a range of psychiatric problems which seeks to calm thoughts by redirecting mental focus through meditative distancing. The mindfulness condition is a non-specific cognitive control for any confounding effect of mood change on symptom relief. CBT follows an 'appraisal' model either through restructuring appraisals and beliefs about the obsession or by de-dramatizing anxious expectations through exposure and reality testing (combined with E/RP). IBT seeks to change the reasoning leading up to the initial inference of doubt on the principle that eliminating the doubt logically and necessarily eliminates all anticipated consequences and accompanying obsessional anxiety. All three treatments will be manualized and administered by experienced professional therapists supervised by a co-investigator with an allegiance to one of the three approaches. The three treatment models operate on distinct processes and on separable stages of the obsessional chain, so therapy components will not overlap. The principal sites chosen will be Montreal Louis-H. Lafontaine Hospital and Gatineau Pierre-Janet Hospital. A total of 80 participants will be recruited over a five-year period into each treatment modality, giving a total of 240, which will permit robust conclusions even with weak effect sizes. Outcome evaluators will be blind to treatment modality and independent of therapists. All therapy will be delivered on an individual weekly basis until significant clinical improvement or up to a maximum of 26 weeks with a 6-month follow-up post-treatment. All parameters of treatment delivery will be identical across treatments. All sessions will be audio recorded and treatment integrity will be rated independently. Outcome measures will be standard DSM-IV based clinical diagnostic scales and also psychosocial measures of end-point functioning across life domains. Treatment process variables will be continuously monitored. Refusal and attrition are calculated at 16% and analysis will include intention to treat. The hypotheses are that: (1) all treatments will be effective in improving mood and reducing symptoms; (2) the IBT will be superior in terms of: (a) its consistent impact over all types of OCD; (b) its lower rate of relapse. The RCT will be the first of its kind in comparing these three active treatments and will impact on treatment of choice for OCD.

ELIGIBILITY:
Inclusion Criteria:

* primary diagnosis according to DSM-IV-TR criteria of OCD
* willingness to keep medication stable while participating in study
* willingness to undergo active psychological treatment
* willingness to undergo randomization into treatment modality
* fluency in either English or French.
* entry criteria do not exclude a secondary diagnosis on Axis I or II providing it does not require treatment or is deemed unlikely to significantly affect compliance with the current treatment plan.
* participants will also be screened on a brief battery of neuropsychological tests to ensure comparability of mental capacity between groups.
* no change in medication type or dose during the 12 weeks before treatment for antidepressants (4 weeks for anxiolytics. If antidepressant or medication as not been stable for at least 12 weeks, a stabilization period will be imposed. Other medication (e.g., anxiolytics) will have to be stable for at least four weeks.

Exclusion Criteria:

* presence of other principal axes 1 disorders requiring treatment
* evidence of suicidal intent
* evidence of current substance abuse
* evidence of current or past of suicidal intent
* evidence of current or past schizophrenia, bipolar disorder or organic mental disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2012-09; Primary Completion 2019-08 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) | Baseline, change after 26 weeks of treatment, change after 6-month follow-up
  The Yale-Brown Obsessive-Compulsive Scale (translation) is the instrument of choice to assess obsessive compulsive symptoms and severity.

SECONDARY OUTCOMES:
Vancouver Obsessional Compulsive Inventory (VOCI) | Baseline, change after 26 weeks of treatment, change after 6-month follow-up
  The Vancouver Obsessional Compulsive Inventory (VOCI)(Translation) to assess a broad spectrum of OCD symptoms and associated personality characteristics.It is a 55-item self-report measure to assess a broad spectrum of OCD symptoms and associated personality characteristics.
Obsessive Beliefs Questionnaire (OBQ-44) | Baseline, change after 26 weeks of treatment, change after 6-month follow-up
  The Obsessive Beliefs Questionnaire (OBQ-44) is a 44-item measure developed by the Obsessive Compulsive Cognitions Working Group between 1995 and 1998. The OBQ consist in three twinned domains based on the working group consensus (over-responsibility/over-estimation of threat, intolerance of uncertainty/over-importance of thought, control of thoughts/perfectionism).
Beck Depression Inventory (BDI) | Baseline, change after 26 weeks of treatment, change after 6-month follow-up
  The Beck Depression Inventory (BDI) (Translation) is a standard 21-item measure to assess depressive symptoms.
Beck Anxiety Inventory (BAI) | Baseline, change after 26 weeks of treatment, change after 6-month follow-up
  The Beck Anxiety Inventory (BAI)(Translation) is a standard 21-item anxiety symptom checklist rating anxiety symptom intensity for the last week on a 0-3 scale.
Over-Values Ideas Scale (OVIS) | Baseline, change after 26 weeks of treatment, change after 6-month follow-up
  Over-Valued Ideas Scale (OVIS)(Translation)is a 11-item clinician-rated scale measuring degree of conviction, insight, justification and actions following from belief.
Inferential Confusion Questionnaire (ICQ) | Baseline, change after 26 weeks of treatment, change after 6-month follow-up
  The ICQ was originally developed in French and is a 30-item questionnaire.
Semi-structured interview to assess primary inference process | Baseline, change after 26 weeks of treatment, change after 6-month follow-up
  Primary inference processes will be rated by semi-structured interview for each obsession on a clinical scale, and daily by the participant, in the daily diary. Strength is rated 0-100 in accordance with how probable the participant considers the primary belief whether it is a doubt "maybe the door isn't locked properly".
Mindful Attention Awareness Scale (MAAS) | Baseline, change after 26 weeks of treatment, change after 6-month follow-up
  The MAAS is a 15-item questionnaire which measures the tendency to be attentive and aware of present moment experience in everyday life and does not require extensive experience with mindfulness. It is uni-dimensional and is appropriate for exploring changes in awareness and attention associated with mindfulness-based stress reduction (MBSR) and is predictive of mood and adaptive regulation.
Global Assessment of Functioning (GAF) scale (DSM-IV, Axis V) | Baseline, change after 26 weeks of treatment, change after 6-month follow-up
  The GAF is a standard DSM measure of adaptation and functioning scored from 0-100.
Systematic Quality of Life Inventory | Baseline, change after 26 weeks of treatment, change after 6-month follow-up
  The Systematic Quality of Life Inventory measure 30 life domains, using three subscales: actual state, goal state and the difference between actual and desired goals of quality of life.
Life Experience Survey | Baseline, change after 26 weeks of treatment, change after 6-month follow-up
  The Life Experience Survey measures negative and positive life events and their impact over 57 life domains.
Social Support Questionnaire | Baseline, change after 26 weeks of treatment, change after 6-month follow-up
  The Social Support Questionnaire has two scales measuring amount and degree of satisfaction with social support.
Social Self-esteem Inventory | Baseline, change after 26 weeks of treatment, change after 6-month follow-up
  The Social Self-esteem Inventory measures agreement on 30 self-statements.

OTHER OUTCOMES:
Clinical Interview | pre-treatment, post-treatment and 6 month follow-up
  A clinical interview assesses content, form, and appraisal of obsessions as well as neutralization strategies used with the target obsession.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Aardema, Ph. D., Principal Investigator — Centre de Recherche de l'Institut Universitaire en santé Mentale de Montréal
Locations (1):
- Centre de recherche de l'Institut universitaire en santé mentale de Montréal, Montreal, Quebec, Canada